CLINICAL TRIAL: NCT05548010
Title: Evaluation of a Short Educational Materials in Improving the Knowledge Level of Venous Thromboembolism and the Compliance of Thromboprophylaxis in Post-operative Patients: a Prospective Study
Brief Title: Venous Thromboembolism (VTE) Knowledge
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, GuangMing Tan, Professor, Chinese University of Hong Kong
Other Study IDs: VTE
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Thromboembolism
MeSH Terms: conditions — Thromboembolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects: Patients >18years old with scheduled operation
  Interventions: Other: No intervention as this is an observational study
- Healthcare Professionals (HCP): HCP of the enrolled subjects
  Interventions: Other: No intervention as this is an observational study

INTERVENTIONS:
Other: No intervention as this is an observational study — No intervention

SUMMARY:
Venous thromboembolism (VTE) is common especially among post-operative patients, and its occurrence is associated with significant morbidity and mortality. VTE is highly preventable with prophylactic modalities ranging from conservative measures such as early mobilization, to mechanical prophylaxis such as intermittent pneumatic compression (ICP), to pharmacological prophylaxis such as peri-operative anticoagulation. Despite established guidelines from various professional societies, the practice of VTE prophylaxis varied greatly from institute to institute. Evidence suggests that there is a significant gap between the optimal thromboprophylaxis as suggested by experts and real-work practice. Many healthcare-providers (HCP) and patients at risk of VTE are either not aware of the risk of VTE or not confident to apply the necessary thromboprophylaxis. The knowledge level of VTE appears to play a key role in affecting the level of compliance to the optimal thromboprophylaxis. Considerable improvement in VTE prophylaxis utilization may result from the implementation of a multifaceted educational program. By improving patient's awareness on VTE prophylaxis, the incidence of DVT might be reduced. The knowledge level of patients can be improved by various means including educational video, administrative measures, or continue medical education program. However, no prospective study has been performed to assess the impact of an educational program on the VTE knowledge level among post-operative patients and their HCP, and if any improvement of their knowledge level can be translated to a better adherence to VTE prophylaxis guidelines. We therefore propose to conduct a prospective non-randomized controlled study to evaluate the effect of an education materials for the patients as well as their HCP on their knowledge level as well as the utilization and adherence of VTE prophylaxis in these patients by comparing two groups of patients and HCP.

ELIGIBILITY:
Inclusion Criteria:

* Capable of providing written informed consent and willing and able to adhere to all protocol requirements
* Male or female at least 18 years of age at the time of providing written informed consent
* Adult patients age >18 scheduled for surgical operations
* Healthcare Providers directedly involve in patients care of these surgical patients.

Exclusion criteria

* Unable to make their own informed consent
* Unable to understand the study protocol
* Visually or auditorily impaired.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The first group will be adult patients age >18 scheduled for surgical operations. The second group will be the HCPs directedly involve in patients care of these surgical patients.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2024-08-04 (Actual)

PRIMARY OUTCOMES:
Difference in VTE knowledge between 2 groups | 4 weeks
  Difference between the knowledge level in the subject group and HCP group after the administration of the educational materials as measured with questionnaire
VTE prophylaxis prescription by healthcare providers | 4 weeks
  Difference in VTE prophylaxis prescribed by HCP after the administration of the educational materials assessed upon patient follow-up/ discharge as reflected by drug prescription sheet and discharge summary
VTE prophylaxis adherence | 4 weeks
  VTE prophylaxis will be advised to subjects upon discharge. Difference in VTE prophylaxis adherence of subjects after the administration of the educational materials will be assessed verbally during follow-up consultation by investigators.

SECONDARY OUTCOMES:
Difference in VTE knowledge level within the HCP group | 4 weeks
  difference in VTE knowledge level within the HCP group before and after the administration of the educational materials as measured with questionnaire.
Difference in patient satisfaction | 4 weeks
  Difference in patient satisfaction scoring before and after the administration of the educational materials to the HCPs assessed during patient follow-up consultation by investigators
Difference in the rate of venous thromboembolism (VTE) | 4 weeks
  Difference in rate of VTE in the HCP group before and after the administration of the educational materials.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Yan, Study Chair — Chinese University of Hong Kong; Guangming Tan, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong